CLINICAL TRIAL: NCT01997957
Title: A Randomized Controled Trial of Oral S-1 in Combination With Sequential Hepatic Arterial Infusion of Oxaliplatin After Transarterial Chemoembolization in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A RCT of Oral S-1 in Combination With Sequential HAIC of Oxaliplatin After TACE in Patients With Advanced HCC
Acronym: SOON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Xu (Other)
Responsible Party: Sponsor-Investigator, Zhu Xu, Interventional Therapy Department, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_06366
Record Dates: First submitted 2013-11-20; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial Chemoembolization; Hepatic Arterial Infusion Chemotherapy; Efficacy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TACE+HAIC-OXA+S-1 (Experimental)
  Interventions: Drug: S-1
- TACE+HAIC-OXA (No Intervention)

INTERVENTIONS:
Drug: S-1 — Begin oral administration of S-1 from the 2nd day after TACE therapy plus arterial indwelling catheter chemotherapy (Oxaliplatin)
  Arms: TACE+HAIC-OXA+S-1

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most commonly malignant tumors around the world and causes death of about 600000~1000000 people each year. Since 1990s, hepatic carcinoma has become the second carcinoma killer in China. Surgical resection or liver transplantation is the only method possibly able to cure hepatic carcinoma. However, due to multiple tumors or poor hepatic function reserve in cirrhosis, surgical treatment is suitable for only a small portion of patients (11.9%-30.1%). Therefore, in clinical practice, transarterial chemoembolization (TACE) or transarterial embolization (TAE) is a preferential and standard treatment of unresectable advanced hepatic carcinoma and has notable advantages in controlling local tumors of the liver. Hepatic arterial infusion of oxaliplatin after TACE can significantly increase the local doses of chemotherapeutic agents in the liver, kill micrometastases and residual foci after embolization and demonstrate outstanding efficacy for treating concomitant portal and hepatic vein tumor thrombi. S-1 is a chemotherapeutic agent with convenient use and definite efficacy and, when used concomitantly with TACE, theoretically can not only effectively control intrahepatic foci but also prevent and control extrahepatic metastatic foci. However, this hasn't been verified in clinical application. This study is intended to investigate efficacy and safety of the combination treatment so as to provide a more effective and safety way for treating patients with advanced hepatic carcinoma (Barcelona stage-C patients with concomitant portal vein tumor thrombi or extrahepatic metastasis).

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form;
* Diagnosed with HCC

Patients with hepatic cirrhosis must comply with AASLD (American Association for the Study of Liver Diseases) diagnostic criteria:

Typical radiological examination (ultrasonography, CT or MRI) manifestations: dynamic enhanced examination shows arterial-phase rapid heterogeneous enhancement and reduced venous-phase or delayed-phase rapid enhancement of space occupation in liver;

* If the diameter of space occupation in liver is ≥2cm, the diagnosis can be established if any of radiological examinations shows the above HCC characteristics;
* If the diameter of space occupation in liver is 1-2cm, the diagnosis can be established only when two radiological examinations show the above HCC characteristics;
* If the diameter of space occupation in liver is≤1cm, histopathological examination is needed for establishing the diagnosis.

Histopathological examination is needed for establishing the diagnosis for patients without hepatic cirrhosis.

* Stage Barcelona C
* Grade A or B Child-Pugh score
* ECOG PS score is 0-1
* At least one measurable focus in liver according to (M) RECIST 1.0 criteria
* Male or female, age>18
* Can orally take drugs
* Anticipated survival≥12 weeks
* Pregnancy test of women at child-bearing ages must be negative within the 7 days before treatment
* Male or female patients included must take effective contraceptive measures during the study period and within 4 weeks after completion of the study
* Within the 7 days before inclusion, bone marrow, liver and kidney functions must satisfy the following requirements:

  * Hemoglobin≥ 90 g/L
  * Absolute neutrophil count (ANC) >1,500/mm3
  * Platelet count≥ 80x109/L
  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 times the upper normal limit (UNL)
  * Total bilirubin < 3UNL
  * Alkaline phosphatase < 4UNL
  * Serum creatinine < 1.5 UNL
  * Amylase and lipase < 2 UNL
  * INR<2.3 or PPT< 1.5 UNL (Patients who are accepting Warfarin or heparin anticoagulant therapy may be included if no evidence is available proving the above indicators are abnormal, but intense monitoring must be exercised. Tests shall be carried out at least once per week until stable INR.)

Exclusion Criteria:

* Early or middle-stage primary HCC
* Any contraindication of TACE therapy

  * Known hepatofugal blood flow
  * Known portal-systemic shunt
  * Abnormal coagulation test (PLT<6000/mm3, thrombogen activity<50%)
  * Renal failure or renal insufficiency necessitating dialysis
  * Serious atherosclerosis
* Foci having undergone local treatment (e.g. resection, RFA, PEI or argon-helium cryoablation) cannot be used as the target foci
* Local therapy or systemic chemotherapy within 4 weeks before inclusion or during the study period
* Acute toxic reaction of CTC grade AE2 or above in any local treatment before inclusion
* History of heart diseases:

  * Congestive heart failure of NYHA grade 2 above
  * Symptomatic coronary artery disease
  * Arrhythmia needing treatment with β blockers or drugs other than digoxin
  * uncontrollable hypertension
* HIV infection or AIDS-related diseases
* Serious active infections other than hepatitis B and hepatitis C (NCI-CTCAE 4.0 grade 2 above)
* Gastrointestinal hemorrhage event within 4 weeks before inclusion
* Thrombogenesis or embolism event within 6 months before inclusion, e.g. cerebral vascular accidents (including TIA), deep venous thrombogenesis or pulmonary embolisms
* Past or present history of concomitant tumors completely different from HCC in primary lesions or histology, excluding head and neck carcinoma in situ, cured basal cell carcinoma, superficial bladder carcinoma (Ta, Tis, T1) and tumors having been cured 3 years before inclusion
* Drug abuse, or psychological or mental diseases that may interfere with the study compliance
* Known or suspected allergy to the study drug or concomitant medications
* Contraindications of S-1
* Pregnancy or lactation
* Any disease that may affect evaluation of the study drug
* Any instability or condition that may impair the patient's safety and compliance in the study
* Gastrointestinal diseases affecting absorption or pharmacokinetics
* Conditions restricting the patient from taking drugs orally, including serious upper gastrointestinal obstruction
* Having accepted TACE before inclusion
* Having taken S-1 before inclusion
* Having accepted liver radiotherapy before inclusion or during the study period
* Having accepted biological regulators, e.g. G-CSF, within the 3 weeks before inclusion
* Having accepted autologous bone marrow transplantation or stem cell transplantation within 1 year before inclusion
* History of homoplastic transplantation
* Any drug that may affect absorption or pharmacokinetics of the study drug
* Poor compliance considered by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Time to progression(TTP) | Up to 2 years
  Time to clinically definite disease progression

SECONDARY OUTCOMES:
Overall survival(OS) | Up to 2 years
Response rate (RR) | Up to 2 years
  The percentage of patients showing partial or complete response to the given treatment
Disease Control Rate (DCR) | Up to 2 years
  The percentage of patients showing partial or complete response or stable disease to the given treatment
Number of Participants with Serious and Non-Serious Adverse Events | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Xu, Master, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China